CLINICAL TRIAL: NCT02455466
Title: Altered PSA Test Due to Possible Suspected Heterophilic Antibodies
Status: Terminated | Type: Observational
Why Stopped: not enough recruitment
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-0652
Record Dates: First submitted 2015-05-11; First posted 2015-05-27 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: PSA

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum of patients
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate if clinically non explainable high or low Prostate-specific antigen (PSA) levels are associated with heterophilic antibodies in the serum of participants. The investigators will examine if heterophilic antibodies are the reasons of altered PSA levels.

ELIGIBILITY:
Inclusion Criteria:

* Male, with a a clinically high or low unexplainable PSA measurement
* Age between 40 and 90 years
* Written informed consent

Exclusion Criteria:

* Female
* No PSA measurement available or planned
* Age over 90 or under 40 years

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male, where a PSA measurement is planned
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Presence of heterophilic antibodies in the serum of participants | 1.5 years
  Heterophilic antibodies will be measured in the Blood serum of participants by sandwich Elisa assay
Altered PSA levels due to the Presence of Heterophilic antibodies | 1.5 years
  If heterophilic antibodies were present in the serum of the participant, another PSA test will be ran after absorbance of heterophilic antibodies to investigate whether PSA levels are changed without the presence of heterophilic antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zürich, Zurich, Switzerland